CLINICAL TRIAL: NCT05145114
Title: Hemodynamic Repercussions in Different Therapeutic Positions in Premature Newborn Under Invasive Mechanical Ventilation
Brief Title: Hemodynamic Repercussions in Different Therapeutic Positions in Premature Newborn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amazon University (Other)
Responsible Party: Principal Investigator, Paulo Eduardo Santos Avila, Principal Investigator, Amazon University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 3.983.789
Record Dates: First submitted 2021-10-04; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Therapeutic Position; Hemodynamics
Keywords: Premature newborn; Patient Positioning; Mechanical ventilation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supine Group (SG) (Experimental)
  Interventions: Procedure: THERAPEUTIC POSITIONS
- Prone Group (PG) (Experimental)
  Interventions: Procedure: THERAPEUTIC POSITIONS
- Lateral Decubitus Group (LDG) (Experimental)
  Interventions: Procedure: THERAPEUTIC POSITIONS

INTERVENTIONS:
Procedure: THERAPEUTIC POSITIONS — Therapeutic positioning includes placing infants in prone (prone), supine, side (lateral) decubitus, using restraint devices to provide support, reassurance and physiological stability.

SUMMARY:
Introduction: Prematurity refers to babies born before 37 weeks of gestation that through technological advances survival is increasing, since most of them are referred to the Neonatal Intensive Care Unit (NICU). Hemodynamic monitoring is of fundamental importance in the care provided to critically ill patients and mechanical ventilation (MV) is often used for the recovery and maintenance of newborns, especially premature infants with any pathology that causes cardiorespiratory failure. Considering this, it is necessary to look for ways to treat these newborns (NB), being the therapeutic positioning one of the simplest and most fundamental to reduce the consequences of the mechanical advantages of the respiratory system of newborns. Objective: To evaluate the hemodynamic repercussions in the various therapeutic positions in premature newborns under invasive mechanical ventilation. Method: A field study to be conducted will be randomized on an experimental, quantitative and descriptive character. It will be developed at the Santa Casa de Misericórdia do Pará Foundation (FSCMPa), in the Neonatal Intensive Care Unit. The population to be evaluated will be preterm infants with gestational age ≤37 weeks, on invasive mechanical ventilation, with no congenital malformations, with the diagnosis of intracranial hemorrhage and that those responsible, after being informed, authorized to participate in the research. Being excluded the preterm infants without legal companion, who are affected by any unfavorable clinical condition, which makes the change of unfeasible position, children with neuromuscular diseases, tracheostomized. A sample will be randomly selected in groups: Prono Group (GP), Supine Group (GS) and Lateral Decubitus Group (GDL). The decubitus to be adopted for each research subject will then be registered by the researcher in a specific form, recording as respiratory cardiological responses: respiratory rate (RR), heart rate (HR) and peripheral oxygen saturation (SPO2), temperature (T) and pressure blood pressure (BP). Such clinical responses will be noted prior to NB positioning, then positioned according to the group to which they will belong for 30 minutes, and then there will be another selection of vital signs.

DETAILED DESCRIPTION:
The present field study to be carried out will be controlled clinical trial, randomized, experimental, quantitative and analytical. The research will be carried out in accordance with the ethical aspects recommended in the Declaration of Helsinki and Nuremberg Code, and by the research standards that may involve human beings of the National Health Council. Parents and guardians of premature newborns eligible for the survey will be invited to consent to the participation of newborns in the survey, in which the purpose, objectives and procedures of the research will be explained, requesting the signature of the Informed Consent Form and Informed and the Informed Consent Term.Then, access to data related to the newborn's medical record will be performed through the presentation of the Data Use Commitment Term. The sample will be randomly separated into groups: Prone Group, Supine Group and Lateral Decubitus Group. The decubitus to be adopted for each research subject will then be registered by the researcher in a specific form that will contain the following information: identification, gender, Apgar in the first and fifth minutes, GA, weight, use of surfactant and amount of doses, time of use of mechanical ventilation, length of hospital stay and others, with this information being obtained from the newborn's medical record, this step will provide data that will characterize the sample. For data acquisition via medical records, the researcher will submit the consent form for data use. The most used physiological parameters are vital signs, such as heart rate and percutaneous oxygen saturation, as they are the most easily observed responses. The most used physiological parameters are vital signs, such as heart rate and percutaneous oxygen saturation, as they are the most easily observed responses. This is due to the fact that babies who need intensive care are usually under these assessments constantly by pulse oximeters and because they have been the best scientifically validated among the physiological responses. The vital signs of heart rate (HR), often respiratory rate (RR) and blood pressure (BP), can be influenced by the infant 's age and health condition. Peripheral oxygen saturation may have its results altered by the baby's behavioral state and pulmonary conditions. The assessment of HR and RR, indirectly, may reflect respiratory discomfort, it is common to observe tachypnea and some patients present tachycardia for not accepting or tolerating the positioning they are submitted. To record the monitoring of cardiorespiratory physiological responses, an interval of 2 hours after the diet will be respected so that there are no complications during the procedure. The respiratory rate (RR) will be collected for this, the thoracic incursions of the patients will be observed for one minute, counted on a digital clock, and to measure the heart rate (HR) and peripheral oxygen saturation, a pulse oximeter will be used, provided by the institution , positioned on the newborn's foot. Axillary temperature will also be measured with a thermometer specific to each NB and blood pressure with a device from the institution.

Such clinical responses will be noted before the positioning of the NB, then participants will be positioned according to the group they belong to for 30 minutes, and then there will be a new verification of vital signs. During the time they are positioned, the RN will be asked not to receive routine procedures from the NICU or any stimulation by the health team. Only in cases that require urgent intervention. Being evaluated 1 times a day in the morning shift for two weeks. The collected data will be stored in Microsoft Excel® spreadsheets , which will serve to perform a simple descriptive statistics that will be presented in percentages, arranged in graphs and tables. Statistical analysis will be based on the use of statistical tests that best fit the study proposal through the Biostat ® statistical package . In order to know the profile of the data, the Shapiro-Wilk test will be applied to verify whether the data under analysis presented normality. To compare the mean values of the data, the ANOVA test will be performed, followed by the Newman-Keuls multiple comparison test for the variables: heart rate, respiratory rate, oxygen saturation and the Studen t test for the variables: blood pressure and axillary temperature. In all tests, the level for rejecting the null hypothesis will be set at 5% (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

* PTNB with GA ≤37 weeks
* In ventilation invasive mechanics
* With absence of congenital malformations
* With absence a diagnosis of intracranial hemorrhage
* That the guardians after being informed, authorized to participate in the research

Exclusion Criteria:

* PTNB without a legal companion
* Who are affected by some unfavorable clinical condition that makes it impossible to change position
* Children with neuromuscular diseases
* Tracheostomized

Ages: 1 Day to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Vital sign of respiratory rate (rpm) will be measured before and after in different therapeutic positions of premature newborns under invasive mechanical ventilation. | Each newborn will be evaluated for only two weeks, being evaluated once a day, in the morning shift.
  The respiratory rate (irpm) will be checked on the mechanical ventilator, noted before the positioning of premature newborns. Next, the newborns will be positioned according to the group and then there will be a recheck of the respiratory rate.
Heart rate vital sign (bpm) will be measured before and after at different therapeutic positions of premature newborns under invasive mechanical ventilation. | Each newborn will be evaluated for only two weeks, being evaluated once a day, in the morning shift.
  The heart rate (bpm) will be checked on the multiparametric vital signs monitor with a value verified by means of electrodes adhered to the patients' chest, noted before the positioning of the premature newborns. Next, the newborns will be positioned according to the group and then there will be a new heart rate check.
Vital sign of peripheral oxygen saturation (percentage) will be measured before and after in different therapeutic positions of premature newborns under invasive mechanical ventilation. | Each newborn will be evaluated for only two weeks, being evaluated once a day, in the morning shift.
  Peripheral oxygen saturation (percentage) will be verified in the multiparametric vital signs monitor with a value verified through the finger oximeter, noted before the positioning of the premature newborns. Next, the newborns will be positioned according to the group and then there will be a new check for peripheral oxygen saturation.
Vital sign of temperature (degree Celsius) will be measured before and after in different therapeutic positions of preterm newborns under invasive mechanical ventilation. | Each newborn will be evaluated for only two weeks, being evaluated once a day, in the morning shift.
  The temperature (degree Celsius) will be checked in the multiparametric vital signs monitor with a value verified by means of a sensor attached to the patient's axillary region, noted before the positioning of the premature newborns. Next, the newborns will be positioned according to the group they and then there will be a new temperature check.
Blood pressure vital sign (mmHg) will be measured before and afterat different therapeutic positions of premature newborns under invasive mechanical ventilation. | Each newborn will be evaluated for only two weeks, being evaluated once a day, in the morning shift.
  Blood pressure (mmHg) will be checked on the multiparametric vital signs monitor with a value verified by means of a pressure cuff placed on the patient's upper limb, noted before the positioning of the premature newborns. Next, the newborns will be positioned according to the group and then there will be a new blood pressure check.

CONTACTS AND LOCATIONS:
Locations (1):
- Paulo Eduardo Santos Avila, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DE CARVALHO MORSCH, A. L. B. et al. Análise das repercussões clínicas da aplicação da posição prona em prematuros sem doença pulmonar. ERSPECTIVA, Erechim. v. 42, Edição Especial, p. 07-14, março, 2018.
- [Background] DE CORDOBA LANZA, F.; BARCELLOS, P.G.; DAL CORSO, S. Benefícios do decúbito ventral associado ao CPAP em recém-nascidos prematuros. Fisioterapia e Pesquisa, v. 19, n. 2, p. 135-140, 2012.
- [Background] DE SÁ, F. E. et al. Estudo sobre os efeitos fisiológicos da técnica de aumento do fluxo expiratório lento em prematuros. Fisioterapia & Saúde Funcional, v. 1, n. 1, p. 16-21, 2012.
- [Background] Oliveira TG, Rego MA, Pereira NC, Vaz LO, Franca DC, Vieira DS, Parreira VF. Prone position and reduced thoracoabdominal asynchrony in preterm newborns. J Pediatr (Rio J). 2009 Sep-Oct;85(5):443-8. doi: 10.2223/JPED.1932. English, Portuguese. PMID 19830358
- [Background] Ramada NC, Almeida Fde A, Cunha ML. Therapeutic touch: influence on vital signs of newborns. Einstein (Sao Paulo). 2013 Dec;11(4):421-5. doi: 10.1590/s1679-45082013000400003. PMID 24488378
- [Result] Hough JL, Johnston L, Brauer SG, Woodgate PG, Pham TM, Schibler A. Effect of body position on ventilation distribution in preterm infants on continuous positive airway pressure. Pediatr Crit Care Med. 2012 Jul;13(4):446-51. doi: 10.1097/PCC.0b013e31822f18d9. PMID 21926660